CLINICAL TRIAL: NCT06622603
Title: A Prospective, Multicenter, Randomized Investigator Initiative Clinical Trial Study on the Effects of Febuxostat Dose Tapering in Gout Patients Optimally Controlled for 5 Years or More
Brief Title: The Effects of Febuxostat Dose Tapering in Gout Patients Optimally Controlled for 5 Years or More
Acronym: TARGET
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Gachon University Gil Medical Center (Other); SMG-SNU Boramae Medical Center (Other); Chungnam National University Hospital (Other); Seoul National University Bundang Hospital (Other); Eulji University Hospital (Other); Ajou University Medical Center (Unknown)
Responsible Party: Principal Investigator, Yun Jong Lee, Professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TARGET-V1-01
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-07

CONDITIONS: Gout; Uric Acid
Keywords: Febuxostat; Allopurinol
MeSH Terms: conditions — Gout | interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Discontinuing group (Placebo Comparator): They (n=15) will take a placebo once daily for 6 months, followed by febuxostat 20 mg once daily for the next 6 months. Randomization is stratified based on the urinary urate excretion rate (≤5.5% vs. >5.5%).
  Interventions: Drug: Febuxostat
- Reducing group (Active Comparator): They (n=29) will take febuxostat 20 mg once daily for 12 months. Randomization is stratified based on the urinary urate excretion rate (≤5.5% vs. >5.5%).
  Interventions: Drug: Febuxostat
- Maintaining group (No Intervention): To serve as an observational reference group, they (n=15) will continue their urate-lowering agents for 12 months. Randomization is stratified based on the urinary urate excretion rate (≤5.5% vs. >5.5%).

INTERVENTIONS:
Drug: Febuxostat — The minimal approved dose of febuxostat is 40 mg/day. We will use 0.5 tablet of febuxostat 40 mg or its placebo.
  Other Names: Usoric® Tab 40mg
  Arms: Discontinuing group; Reducing group

SUMMARY:
The goal of this clinical trial is to compare the changes in serum urate levels and symptom recurrence after reducing or suspending urate-lowering agents in well-controlled gout patients (the 'after dishes are clean' state in the Dirty Dish hypothesis)

Researchers will compare three randomized groups: the reducing group takes febuxostat 20 mg once daily for 12 months, the discontinuing group takes a placebo once daily for 6 months, followed by febuxostat 20 mg once daily for the next 6 months, and the maintaining group continues their pre-study urate-lowering agents for 12 months, serving as an observational reference group.

During the 12-month study period, participants will visit every 3 months for laboratory evaluations including serum urate levels, and for checking symptomatic status using questionnaires and diaries. Additionally, musculoskeletal ultrasonography and serum sample collection will be performed at baseline to study predictors for maintaining serum urate levels <7.0 mg/dL after reducing or suspending urate-lowering therapy.

DETAILED DESCRIPTION:
1. Background

1. Hyperuricemia is a condition that underlies the development of gout. Gout incidence has been reported as 1.1% with urate levels <6 mg/dL and 3% with urate levels between 6-7 mg/dL in longitudinal studies. However, few studies have examined the incidence after suspending urate-lowering therapy following long-term maintenance of serum urate <6 mg/dL.
2. A US study found that gout patients who maintained serum urate <6.0 mg/dL for over 5 years and had resolved tophi did not experience flare-ups if levels remained <7 mg/dL, while recurrence occurred in those with levels >7 mg/dL. Based on these findings, the study proposed a two-stage gout treatment strategy, known as the "dirty dish" hypothesis.
3. The approved minimum dose of febuxostat is 40 mg/day. Previous studies observed that febuxostat 20 mg/day reduced serum urate levels to <7.0 mg/dL, although it did not meet the current treatment goal during the initial phase.
4. Therefore, a low dose of febuxostat at 20 mg/day could be sufficient to meet the preventive treatment goal of <7 mg/dL proposed by the "dirty dish" hypothesis

2. Sample size determination

1. Average serum urate levels and standard deviations were extracted from 2 previous clinical trials for febuxostat (including 20 mg/day dose) and 3 observational studies on the effects of complete discontinuation of urate-lowering agents. The proportion of patients with serum uric acid levels <7.0 mg/dL was calculated using the normal distribution curve.
2. Based on previous studies, we assumed that the smallest proportion of subjects with serum urate <7.0 mg/dL is 5% for the discontinuing group and 56% for the reducing group. Fisher's exact test (1-β = 0.80, α = 0.05, 2:1 ratio) indicates that 12 subjects are needed for the discontinuing group and 24 for the reducing group. Adjusting for a 15% dropout rate, the final numbers are 15 and 29, respectively.
3. The urate-lowering therapy-maintaining group is expected to have a 100% rate of serum urate <7.0 mg/dL as they are treated according to current guidelines. Therefore, in the case of the maintaining group, 15 subjects - half the number in the discontinuing group - will be assigned to this group without statistical calculation.

2. General principles of statistical analysis

1) Categorical variables will be presented as frequencies and percentages, with 95% CIs if needed. Chi-square tests and Fisher's exact tests will be used for categorical outcomes. For missing data or withdrawals, the analysis will use available data, replacing missing values with the previous measurement.

2) Analysis population

1. SAS (Safety Analysis Set): Includes all participants who received at least one dose of the investigational drug. Safety data analysis will be conducted using SPSS or R.
2. FAS (Full Analysis Set or Intention-to-Treat Set): Includes participants who received at least one dose of the drug and have available primary outcome data (serum urate levels) before and after treatment.
3. PPS (Per-Protocol Set): Consists of FAS participants with no major protocol violations, such as significant inclusion/exclusion criteria breaches, prohibited medication use, or adherence issues. Efficacy analysis will be primarily conducted with the PPS, with additional analysis in the FAS.

3) Efficacy analysis The primary analysis population is the PPS, with sensitivity analysis conducted in the FAS.

4) Safety analysis The primary analysis population is the SAS. Descriptive statistics will be presented and analyzed for all adverse events occurring after the administration of the investigational drug, as well as for clinical laboratory results, vital signs, physical examinations, electrocardiograms, and liver function tests.

ELIGIBILITY:
* Inclusion Criteria:

  1. Adult gout patients aged ≥19 but <80 years.
  2. Gout patients treated with urate-lowering therapy (either allopurinol or febuxostat monotherapy, or a combination of two agents) for at least the past 5 years.
  3. Patients who have at least five serum urate level measurements over the past 5 years and meet one of the following criteria:

     All serum urate levels measured in the past 5 years have been maintained below 6.0 mg/dL; or the area under the curve (AUC) of serum urate levels over time for the past 5 years is less than 33.0 mg/dL x year
  4. Patients without palpable or visible tophi on physical examination (evaluated at pre-defined 18 joint sites and the ears).
  5. Patients without acute gouty attack or history of nephrolithiasis in the past 12 months
  6. Patients with an estimated glomerular filtration rate (eGFR) of 60 mL/min/1.73m² or higher, based on the Cockcroft-Gault formula.
  7. Patients who voluntarily provide written informed consent to participate.
* Exclusion Criteria:

  1. Subjects who continuously require prophylactic low-dose colchicine/NSAIDs.
  2. Subjects already having taken low-dose urate-lowering agents. The low-dose urate-lowering agents are defined as allopurinol ≤200 mg/day or febuxostat ≤20 mg/day. But patients on a combination of low-dose allopurinol and febuxostat are eligible.
  3. Subjects taking medications that could affect serum uric acid levels and uric acid fractional excretion rates, such as benzbromarone, fenofibrate, loop diuretics, thiazide or thiazide-like diuretics, and losartan.
  4. Subjects classified as having high-risk alcohol use according to the National Institute on Alcohol Abuse and Alcoholism (NIAAA):

     For men <65 years: more than 14 drinks per week or for men ≥65 years or women: more than 7 drinks per week
  5. Subjects with a history of hypersensitivity to febuxostat or allopurinol
  6. Subjects with unstable cardiovascular conditions, who require adjustment of urgent their therapy
  7. Subjects taking mercaptopurine or azathioprine
  8. Subjects with genetic issues such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
  9. Subjects with moderate or severe liver dysfunction (AST or ALT levels greater than 3 times the upper normal limit)
  10. Subjects for whom investigators anticipate that a change in a urate-lowering agent dose could present significant risks or that any factor could severely impact drug adherence, complicating study registration.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-14 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with serum urate levels <7.0 mg/dL | 6 months
  The proportion of patients who maintain serum urate levels <7.0 mg/dL at 6 months after taking febuxostat 20 mg once daily or after suspending urate-lowering agents

SECONDARY OUTCOMES:
The proportion of subjects with serum urate <7.0 mg/dL | 6 months and 12 months
  We will compare among maintaining, reducing, and discontinuing groups at 6 months and between maintaining and reducing groups at 12 months
Serum urate levels | 6 months and 12 months
  We will compare among maintaining, reducing, and discontinuing groups at 6 months and between maintaining and reducing groups at 12 months
Gout Impact Scale (GIS) score using the Korean version | 6 months and 12 months
  We will compare among maintaining, reducing, and discontinuing groups at 6 months and between maintaining and reducing groups at 12 months
Patient's overall assessment of gout using a visual analog scale | 6 months and 12 months
  We will compare among maintaining, reducing, and discontinuing groups at 6 months and between maintaining and reducing groups at 12 months
EuroQol(EQ)-5D score | 6 months and 12 months
  We will compare among maintaining, reducing, and discontinuing groups at 6 months and between maintaining and reducing groups at 12 months
Gout activity score (GAS) | 6 months and 12 months
  GAS is calculated as (0.09 × last 12-month attacks) + [1.01 × square root (serum uric acid)] + [0.34 × VAS patient] + [0.53 × ln (1 + tophi number)] We will compare among maintaining, reducing, and discontinuing groups at 6 months and between maintaining and reducing groups at 12 months.
Drug adherence | 6 months and 12 months
  Adherence is defined as defined as taking 80% or more of the prescribed medication (using by the number of remaining pills). We will compare among maintaining, reducing, and discontinuing groups at 6 months and between maintaining and reducing groups at 12 months.
Incidence rate of acute gouty arthritis | 6 months and 12 months
  We will compare among maintaining, reducing, and discontinuing groups at 6 months and between maintaining and reducing groups at 12 months.
Swollen and tender joint counts of 66/68 joints | 6 months and 12 months
  We will compare among maintaining, reducing, and discontinuing groups at 6 months and between maintaining and reducing groups at 12 months.

OTHER OUTCOMES:
The reliability of the ultrasound scoring system for tophi in gout patients | Baseline
  We will compare the USG scores evaluated by each institution with ones evaluated by an independent review committee.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Jong Lee, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dalbeth N, Phipps-Green A, Frampton C, Neogi T, Taylor WJ, Merriman TR. Relationship between serum urate concentration and clinically evident incident gout: an individual participant data analysis. Ann Rheum Dis. 2018 Jul;77(7):1048-1052. doi: 10.1136/annrheumdis-2017-212288. Epub 2018 Feb 20. PMID 29463518
- [Background] Robinson PC, Frampton C, Phipps-Green A, Neogi T, Stamp L, Taylor W, Merriman TR, Dalbeth N. Longitudinal development of incident gout from low-normal baseline serum urate concentrations: individual participant data analysis. BMC Rheumatol. 2021 Aug 28;5(1):33. doi: 10.1186/s41927-021-00204-4. PMID 34452645
- [Background] FitzGerald JD, Dalbeth N, Mikuls T, Brignardello-Petersen R, Guyatt G, Abeles AM, Gelber AC, Harrold LR, Khanna D, King C, Levy G, Libbey C, Mount D, Pillinger MH, Rosenthal A, Singh JA, Sims JE, Smith BJ, Wenger NS, Bae SS, Danve A, Khanna PP, Kim SC, Lenert A, Poon S, Qasim A, Sehra ST, Sharma TSK, Toprover M, Turgunbaev M, Zeng L, Zhang MA, Turner AS, Neogi T. 2020 American College of Rheumatology Guideline for the Management of Gout. Arthritis Care Res (Hoboken). 2020 Jun;72(6):744-760. doi: 10.1002/acr.24180. Epub 2020 May 11. PMID 32391934
- [Background] Scheepers LEJM, van Onna M, Stehouwer CDA, Singh JA, Arts ICW, Boonen A. Medication adherence among patients with gout: A systematic review and meta-analysis. Semin Arthritis Rheum. 2018 Apr;47(5):689-702. doi: 10.1016/j.semarthrit.2017.09.007. Epub 2017 Oct 7. PMID 29198878
- [Background] Kim A, Kim Y, Kim GT, Ahn E, So MW, Lee SG. Comparison of persistence rates between allopurinol and febuxostat as first-line urate-lowering therapy in patients with gout: an 8-year retrospective cohort study. Clin Rheumatol. 2020 Dec;39(12):3769-3776. doi: 10.1007/s10067-020-05161-w. Epub 2020 May 26. PMID 32458236
- [Background] Perez-Ruiz F, Herrero-Beites AM, Carmona L. A two-stage approach to the treatment of hyperuricemia in gout: the "dirty dish" hypothesis. Arthritis Rheum. 2011 Dec;63(12):4002-6. doi: 10.1002/art.30649. PMID 21898351
- [Background] Loebl WY, Scott JT. Withdrawal of allopurinol in patients with gout. Ann Rheum Dis. 1974 Jul;33(4):304-7. doi: 10.1136/ard.33.4.304. No abstract available. PMID 4416909
- [Background] Perez-Ruiz F, Atxotegi J, Hernando I, Calabozo M, Nolla JM. Using serum urate levels to determine the period free of gouty symptoms after withdrawal of long-term urate-lowering therapy: a prospective study. Arthritis Rheum. 2006 Oct 15;55(5):786-90. doi: 10.1002/art.22232. PMID 17013833
- [Background] Komoriya K, Hoshide S, Takeda K, Kobayashi H, Kubo J, Tsuchimoto M, Nakachi T, Yamanaka H, Kamatani N. Pharmacokinetics and pharmacodynamics of febuxostat (TMX-67), a non-purine selective inhibitor of xanthine oxidase/xanthine dehydrogenase (NPSIXO) in patients with gout and/or hyperuricemia. Nucleosides Nucleotides Nucleic Acids. 2004 Oct;23(8-9):1119-22. doi: 10.1081/NCN-200027381. PMID 15571213
- [Background] Kamatani N, Fujimori S, Hada T, Hosoya T, Kohri K, Nakamura T, Ueda T, Yamamoto T, Yamanaka H, Matsuzawa Y. Placebo-controlled, double-blind study of the non-purine-selective xanthine oxidase inhibitor Febuxostat (TMX-67) in patients with hyperuricemia including those with gout in Japan: phase 3 clinical study. J Clin Rheumatol. 2011 Jun;17(4 Suppl 2):S19-26. doi: 10.1097/RHU.0b013e31821d36de. PMID 21654266
- [Background] Liang N, Sun M, Sun R, Xu T, Cui L, Wang C, Ma L, Cheng X, Xue X, Sun W, Yuan X, Zhang H, Li H, He Y, Ji A, Wu X, Li C. Baseline urate level and renal function predict outcomes of urate-lowering therapy using low doses of febuxostat and benzbromarone: a prospective, randomized controlled study in a Chinese primary gout cohort. Arthritis Res Ther. 2019 Sep 2;21(1):200. doi: 10.1186/s13075-019-1976-x. PMID 31477161
- [Background] Yan F, Xue X, Lu J, Dalbeth N, Qi H, Yu Q, Wang C, Sun M, Cui L, Liu Z, He Y, Yuan X, Chen Y, Cheng X, Ma L, Li H, Ji A, Hu S, Ran Z, Terkeltaub R, Li C. Superiority of Low-Dose Benzbromarone to Low-Dose Febuxostat in a Prospective, Randomized Comparative Effectiveness Trial in Gout Patients With Renal Uric Acid Underexcretion. Arthritis Rheumatol. 2022 Dec;74(12):2015-2023. doi: 10.1002/art.42266. Epub 2022 Nov 11. PMID 35795968
- [Background] Morillon MB, Christensen R, Singh JA, Dalbeth N, Saag K, Taylor WJ, Neogi T, Kennedy MA, Pedersen BM, McCarthy GM, Shea B, Diaz-Torne C, Tedeschi SK, Grainger R, Abhishek A, Gaffo A, Nielsen SM, Noerup A, Simon LS, Lassere M, Tugwell P, Stamp LK, Gout Working Group FTO. Serum urate as a proposed surrogate outcome measure in gout trials: From the OMERACT working group. Semin Arthritis Rheum. 2021 Dec;51(6):1378-1385. doi: 10.1016/j.semarthrit.2021.11.004. Epub 2021 Nov 15. PMID 34839932
- [Background] Khosravan R, Grabowski BA, Wu JT, Joseph-Ridge N, Vernillet L. Pharmacokinetics, pharmacodynamics and safety of febuxostat, a non-purine selective inhibitor of xanthine oxidase, in a dose escalation study in healthy subjects. Clin Pharmacokinet. 2006;45(8):821-41. doi: 10.2165/00003088-200645080-00005. PMID 16884320
- [Background] Hirsch JD, Terkeltaub R, Khanna D, Singh J, Sarkin A, Shieh M, Kavanaugh A, Lee SJ. Gout disease-specific quality of life and the association with gout characteristics. Patient Relat Outcome Meas. 2010 Mar 1;2010:1-8. doi: 10.2147/PROM.S8310. PMID 21686040
- [Background] Scire CA, Carrara G, Viroli C, Cimmino MA, Taylor WJ, Manara M, Govoni M, Salaffi F, Punzi L, Montecucco C, Matucci-Cerinic M, Minisola G; Study Group for the Kick-Off of the Italian Network for Gout Study. Development and First Validation of a Disease Activity Score for Gout. Arthritis Care Res (Hoboken). 2016 Oct;68(10):1530-7. doi: 10.1002/acr.22844. Epub 2016 Sep 6. PMID 26815286
- [Background] La-Crette J, Jenkins W, Fernandes G, Valdes AM, Doherty M, Abhishek A. First validation of the gout activity score against gout impact scale in a primary care based gout cohort. Joint Bone Spine. 2018 May;85(3):323-325. doi: 10.1016/j.jbspin.2017.05.010. Epub 2017 May 17. PMID 28528279
- [Background] Ichida K, Matsuo H, Takada T, Nakayama A, Murakami K, Shimizu T, Yamanashi Y, Kasuga H, Nakashima H, Nakamura T, Takada Y, Kawamura Y, Inoue H, Okada C, Utsumi Y, Ikebuchi Y, Ito K, Nakamura M, Shinohara Y, Hosoyamada M, Sakurai Y, Shinomiya N, Hosoya T, Suzuki H. Decreased extra-renal urate excretion is a common cause of hyperuricemia. Nat Commun. 2012 Apr 3;3:764. doi: 10.1038/ncomms1756. PMID 22473008
- [Background] Gaffo AL, Dalbeth N, Saag KG, Singh JA, Rahn EJ, Mudano AS, Chen YH, Lin CT, Bourke S, Louthrenoo W, Vazquez-Mellado J, Hernandez-Llinas H, Neogi T, Vargas-Santos AB, da Rocha Castelar-Pinheiro G, Amorim RBC, Uhlig T, Hammer HB, Eliseev M, Perez-Ruiz F, Cavagna L, McCarthy GM, Stamp LK, Gerritsen M, Fana V, Sivera F, Taylor W. Brief Report: Validation of a Definition of Flare in Patients With Established Gout. Arthritis Rheumatol. 2018 Mar;70(3):462-467. doi: 10.1002/art.40381. Epub 2018 Feb 6. PMID 29161469
- [Background] Cipolletta E, Di Battista J, Di Carlo M, Di Matteo A, Salaffi F, Grassi W, Filippucci E. Sonographic estimation of monosodium urate burden predicts the fulfillment of the 2016 remission criteria for gout: a 12-month study. Arthritis Res Ther. 2021 Jul 9;23(1):185. doi: 10.1186/s13075-021-02568-x. PMID 34243813
- See also: Gout: diagnosis and management | Guidance - NICE — https://www.nice.org.uk/guidance/ng219/chapter/Recommendations